CLINICAL TRIAL: NCT04181203
Title: An Open Label, Randomized, Phase III Study, Evaluating the Efficacy of a Combination of Apalutamide With Radiotherapy and LHRH Agonist in High-risk Postprostatectomy Biochemically Relapsed Prostate Cancer Patients
Brief Title: Combined Apalutamide, Radiotherapy, and LHRH Agonist in Prostate Cancer Patients After Prostatectomy
Acronym: CARLHA-2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Janssen Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GETUG-AFU33 UC-0160/1702; 2017-000155-21 (EudraCT Number)
Record Dates: First submitted 2019-11-26; First posted 2019-11-29 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
Keywords: Apalutamide; Salvage radiotherapy; Radical prostatectomy; PSA
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; Leuprolide; Goserelin; Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SRT + 6 months of LHRHa (Active Comparator): * Treatment with LHRHa will start 4 weeks before the first RT fraction (i.e Day 1 of Week 1 of treatment period.) The total duration of the LHRHa treatment is 6 months.
  * SRT will start 4 weeks after the first administration of LHRHa (i.e Day 1 of Week 5 of treatment period.). The total duration of SRT is 6.5 weeks.
  Interventions: Radiation: Salvage radiotherapy (SRT); Drug: Luteinising Hormone Releasing Hormone agonist (LHRHa)
- SRT + 6 months of LHRHa + 6 months of Apalutamide (Experimental): * Treatment with LHRHa will start 4 weeks before the first RT fraction (i.e Day 1 of Week 1 of treatment period.) The total duration of the LHRHa treatment is 6 months.
  * Treatment with apalutamide (240 mg PO daily) should start the same day as the first LHRHa administration, for 6 months.
  * SRT will start 4 weeks after the first administration of LHRHa (i.e Day 1 of Week 5 of treatment period.). The total duration of SRT is 6.5 weeks.
  Interventions: Drug: Apalutamide; Radiation: Salvage radiotherapy (SRT); Drug: Luteinising Hormone Releasing Hormone agonist (LHRHa)

INTERVENTIONS:
Drug: Apalutamide — 240 mg PO daily should start the same day as the first LHRHa administration for 6 months.
  months.
  Other Names: ARN-509
  Arms: SRT + 6 months of LHRHa + 6 months of Apalutamide
Radiation: Salvage radiotherapy (SRT) — The SRT treatment will be administered to a total dose of 66 Gy (in 33 fractions of 2 Gy) directed at the prostate bed with an additional 56.1 Gy (in 33 fractions of 1.7 Gy) directed at the pelvis region. The pelvis will be irradiated in all patients.
  An additional simultaneously integrated boost of 69.3 Gy (in 33 fractions of 2.1 Gy) can be delivered to a local relapse based on Positron Emission Tomography - Computed Tomography (PET/CT) and Magnetic Resonance Imaging (MRI) images.
Drug: Luteinising Hormone Releasing Hormone agonist (LHRHa) — Doses of LHRHa may vary due to availability of different brand names and pharmaceutical forms. It will be left to the discretion of the investigator.
  Other Names: leuprolide, goserelin, triptorelin acetate

SUMMARY:
This is a multicenter, randomized, open label, phase III study comparing the efficacy and safety of apatulamide combined with concomitant prostate-bed salvage radiotherapy (SRT) and androgen deprivation therapy (ADT) versus concomitant prostate-bed SRT and ADT in high-risk postprostatectomy biochemically relapsed prostate cancer patients.

DETAILED DESCRIPTION:
The purpose of the CARLHA-2 study is to determine if the combination of apalutamide with 6 months of LHRH agonists and radiotherapy results in an improvement of progression-free survival (PFS) in comparison to the combination of 6 months of LHRH agonists with radiotherapy in high-risk postprostatectomy biochemically relapsed prostate cancer patients.

Radical prostatectomy must have been done at least 6 months before inclusion and is not part of this study.

Patients after radical prostatectomy and biochemical relapse will be randomized in a 1:1 ratio to receive either 6 months of LHRH agonists + SRT or 6 months of LHRH agonists + SRT + 6 months of apalutamide.

The stratification variables include Gleason score, prostate-specific antigen (PSA), negative resection margins, extension to seminal vesicle(s), and PSA doubling time.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have signed a written informed consent form prior to any trial specific procedures
2. Age ≥18 years old and ≤80 years old
3. Histologically confirmed diagnosis of prostate adenocarcinoma treated primarily with radical prostatectomy
4. Tumor stage pT2, pT3 or pT4* (*only in case of bladder neck involvement)
5. Patients should have no clinical and radiological signs (18FCH-PET CT-scan or 68Ga-PSMA-PET CT-scan) of metastatic disease. Patients with a local relapse or pelvic nodal relapse (N1) detected on PET CT-scan can be randomized
6. Eastern Cooperative Oncology Group (ECOG) performance status ≤1
7. PSA ≥0.2 ng/mL at the time of randomization with an elevation of PSA over three consecutive assays. PSA increases over a 1-month interval minimum
8. At least 3 months between radical prostatectomy and randomization.
9. High-risk features as defined by at least one of these characteristics: PSA at relapse >0.5 ng/mL or Gleason score >7 or tumor stage pT3b or resection margins R0 or PSA doubling time ≤6 months or pelvic lymph node relapse (N1, ≤5 lymph nodes)
10. Adequate renal function: serum creatinine <1.5 x upper limit of normal (ULN) or a calculated corrected creatinine clearance ≥60 mL/min according to the Cockcroft-Gault formula, creatinemia <2 ULN
11. Adequate hepatic function: total bilirubin ≤1.5 x ULN (unless documented Gilbert's syndrome), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x ULN
12. Patients with QTc prolongation <500 ms, inclusion should considered after close benefit/risk assessment and cardiologist advice
13. Patients must be willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations
14. Patients must be affiliated to the Social Security System

Exclusion Criteria:

1. Previous treatment with hormone therapy for prostate cancer
2. Histology other than adenocarcinoma
3. Surgical or chemical castration
4. Other malignancy except adequately treated basal cell carcinoma of the skin or other malignancy from which the patient has been cured for at least 5 years
5. Previous pelvic radiotherapy
6. More than 5 (>5) pelvic lymph node relapses
7. Paraaortic, thoracic or supaclavicular nodal relapse (M1a)
8. History of Inflammatory bowel disease or any malabsorption syndrome or conditions that would interfere with enteral absorption
9. Uncontrolled hypertension (defined as systolic blood pressure (BP) ≥140 mmHg or diastolic BP ≥90 mmHg). Patients with a history of hypertension are allowed provided blood pressure is controlled by anti-hypertensive treatment
10. Clinically significant history of liver disease consistent with Child-Pugh class B or C
11. History of seizure or condition that may pre-dispose to seizure (including, but not limited to prior stroke, transient ischemic attack or loss of consciousness ≤1 year prior to randomization; brain arteriovenous malformation or intracranial masses such as schwannomas and meningiomas that are causing edema or mass effect)
12. Medications known to lower the seizure threshold must be discontinued or substituted at least 4 weeks prior to study entry
13. Severe or unstable angina, myocardial infarction, symptomatic congestive heart failure, arterial or venous thromboembolic events (e.g pulmonary embolism, cerebrovascular accident including transient ischemic attacks) or clinically significant ventricular arrhythmias within 6 months prior to randomization
14. Certain risk factors for abnormal heart rhythms/QT prolongation: torsade de pointes ventricular arrhythmias (e.g, heart failure, hypokalemia, or a family history of a long QT syndrome), a QT or corrected QT (QTc) interval >500 ms at baseline
15. Medications known to prolong QTc
16. Known hypersensitivity to apalutamide or to any of its components
17. Galactosemia, Glucose-galactose malabsorption or lactase deficiency
18. Inability or willingness to swallow oral medication
19. Individual deprived of liberty or placed under the authority of a tutor
20. Patients already included in another therapeutic trial with an experimental drug or having been given an experimental drug within the 30 days before inclusion

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Estimated)
Dates: Start 2020-01-09 (Actual); Primary Completion 2028-09-28 (Estimated); Study Completion 2033-12-28 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 5 years
  PFS is defined as the time from the date of randomization to the date of first evidence of loco-regional recurrences, or distant metastases, or death from any cause whichever occurs first, or the date of last known follow-up alive without any such events.

SECONDARY OUTCOMES:
Cancer-specific overall survival | 10 years
  Cancer-specific overall survival is defined as the time from the date of randomization to the date of death related to prostate cancer or the date of last known follow-up alive.
Overall survival (OS) | 10 years
  OS is defined as the time from the date of randomization to the date of death from any cause or the date of last known follow-up alive.
Biochemical relapse-free survival | 10 years
  Biochemical relapse-free survival will be retrospectively defined by the interval between the date of randomization and the date of the first PSA elevation following the 6-months treatment in both arms (PSA ≥0.5 ng/mL confirmed by two consecutive PSA increases over a 2-month interval).
Time to castration resistance | 10 years
  The time to castration resistance is defined as the time from the date of randomization to the date of appearance of castration resistance defined in the European Association of Urology (EAU) guidelines.
Adverse events graded according to the NCI Common Terminology Criteria for Adverse Events version 5.0 | Throughout study completion, up to 10 years
  The NCI Common Terminology Criteria for Adverse Events is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term.
Quality of life questionnaire - Core 30 (QLQ-C30) | At baseline, 3 months, 6 months, every 6 months up to 5 years then every 12 months up to 10 years
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of Life Questionnaire - Prostate Cancer Module (QLQ-PR25) | At baseline, 3 months, 6 months, every 6 months up to 5 years then every 12 months up to 10 years
  This EORTC prostate cancer specific questionnaire is intended to supplement the QLQ-C30.
  The prostate cancer module is a 25-item questionnaire designed for use among patients with localized and metastatic prostate cancer. It includes subscales assessing urinary symptoms (9 items), bowel symptoms (4 items), treatment-related symptoms (6 items) and sexual functioning (6 items). Using a 4-point Likert scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), patients indicate the degree to which they have experienced symptoms.
International Index of Erectile Function (IIEF-5) | At baseline, 3 months, 6 months, every 6 months up to 5 years then every 12 months up to 10 years
  International Index of Erectile Function (IIEF-5) is multidimensional, self-administered questionnaire composed of 15 questions that examine the 4 main domains of male sexual function (erectile function [6 items], orgasmic function [2 items], sexual desire [2 items], and intercourse satisfaction [3 items]) and overall satisfaction (2 items). Using a 6-point Likert scale (questions 1 to 10) and 5-point Likert scale (questions 15 to 15), patients indicate the degree to which they have experienced symptoms. The total score for each domain can therefore classifies the severity of erectile dysfunction into five categories: no (score 26-30), mild (22-25), mild to moderate (17-21), moderate (11-16), and severe (1-10) erectile dysfunction.
Lawton Instrumental Activities of Daily Living (IADL) Scale | At baseline, 3 months, 6 months, every 6 months up to 5 years then every 12 months up to 10 years
  Lawton Instrumental Activities of Daily Living (IADL) Scale is a self-reported questionnaire to assess independent living skills for older adults. This questionnaire, composed of 31 questions organized into 8 domains (ability to use telephone, shopping, food preparation, housekeeping, laundering, mode of transportation, responsibility for own medications, and ability to handle finances), is designed to identify improvement or deterioration of a person functioning over time. Each domain is scored 0-1 for a summary score ranging from 0 (low function, dependent) to 8 (high function, independent).

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane SUPIOT, Principal Investigator — Institut de Cancérologie de l'Ouest - Saint Herblain
Locations (15):
- France (15):
  - Clinique Claude Bernard, Albi
  - Institut de Cancérologie de l'Ouest, Angers
  - Institut Bergonié, Bordeau
  - Centre Georges François LECLERC, Dijon
  - Centre Hospitalier Emile ROUX, Le Puy-en-Velay
  - Centre Oscar Lambret, Lille
  - Institut de Cancérologie de Montpellier, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Institut Jean Godinot, Reims
  - Centre Henri Becquerel, Rouen
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Institut de Cancérologie de la Loire Lucien Neuwirth, Saint-Priest-en-Jarez
  - Institut de Cancérologie Paris Nord, Sarcelles
  - Centre Paul STRAUSS, Strasbourg
  - Clinique Pasteur - ONCORAD, Toulouse

IPD SHARING:
Plan to Share IPD: No